CLINICAL TRIAL: NCT04574193
Title: Continuing Care App for Probationers and Parolees With Substance Use Disorders
Brief Title: Continuing Care App for Probationers and Parolees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: COG Analytics (Other)
Collaborators: Friends Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Steven Carswell, Principal Investigator, COG Analytics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R44MD008848-02 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-10-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The evaluation will involve a two-group RCT in which 100 men and women on probation or parole, who are currently receiving outpatient substance use treatment at THC, will be randomly assigned to one of two conditions: (1) Continuing Care app (CC app; n=50): Participants will receive the CC app, in addition to usual care at the treatment program (12-weeks of weekly group cognitive behavioral therapy), or (2) Treatment As Usual (TAU; n=50): Participants will only receive 12-weeks of weekly group cognitive behavioral therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuing Care App (Experimental): Participants will receive the Continuing Care app, in addition to usual care at the treatment program (12-weeks of weekly group cognitive behavioral therapy).
  Interventions: Device: digital therapeutic for substance use disorders
- Treatment As Usual (Active Comparator): Participants will only receive 12-weeks of weekly group cognitive behavioral therapy.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Device: digital therapeutic for substance use disorders — The Continuing Care application (app) is a HIPAA-compliant, mobile-friendly, software program designed to meet the recovery and personal support needs of probationers and parolees with SUDs who are at elevated risk of relapse, re-arrest, and incarceration.
  Arms: Continuing Care App
Other: Treatment As Usual — 12-weeks of weekly group cognitive behavioral therapy
  Arms: Treatment As Usual

SUMMARY:
This project extends successful Phase I work that developed a Continuing Care mobile application (app) for probationers and parolees with SUDs who are at elevated risk of relapse, re-arrest, and incarceration. This Phase II STTR project will finalize app development and evaluate its efficacy in a randomized controlled trial. The project has high public health significance due to its potential to provide an accessible recovery support tool for individuals on probation or parole that could improve their substance use disorder treatment outcomes.

DETAILED DESCRIPTION:
Substance use disorders (SUDs) continue to be one of the most serious public health problems in the US. Studies have consistently documented a substantially higher prevalence of SUDs among adults under criminal justice supervision in the community (i.e., probation or parole) as compared to the general population. There is growing recognition that addiction is a chronic health condition, and individuals with SUDs typically cycle through multiple periods of treatment, abstinence, and relapse over several years to achieve and maintain recovery. Studies show that continuing care interventions can provide ongoing support or extend primary treatment gains with respect to reducing substance use, relapse, and criminal activity. Recent diffusion of Internet and smartphone technologies among disadvantaged populations now offers unprecedented opportunities for increasing access to quality continuing care interventions as well as chronic disease self-management tools. Probationers and parolees at high risk for drug abuse relapse and involvement in health compromising behaviors are an important population that stands to benefit from continuing care technologies. However, to date, no such technologies exist that are specifically tailored to meet the unique needs of this high-risk population.

Building on our team's extensive experience in the fields of criminology and substance use, we propose to complete the development of a Continuing Care mobile application (app) and conduct a randomized controlled trial to assess efficacy among clients on probation or parole who are enrolled in outpatient substance use treatment. The app is designed to meet the recovery and personal support needs of probationers and parolees with SUDs who are at elevated risk of relapse, re-arrest, and incarceration. It is guided by the principles of the transtheoretical model of behavior change and app content is derived from the Your Own Reintegration System (YOURS) program, an empirically-supported16 intervention that focuses on substance use recovery, reducing criminal thinking and behavior, and managing and building support systems. If proven to be efficacious, the app could be deployed across the national network of outpatient treatment providers, and be highly significant in its direct impact on public health.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently on community supervision (probation or parole) or justice-involvement in the past 12 months
* Currently a client receiving outpatient substance use treatment
* Willing to receive supplemental treatment services through a mobile app
* Willing to provide informed consent and complete research assessments

Exclusion Criteria:

* Severe psychiatric problems (e.g., untreated psychosis, untreated bipolar disorder)
* Suicidality within the past 6-months, as determined by clinical staff, which could make participation in a novel treatment hazardous

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Weeks Retained in Substance Use Treatment | up to 12 weeks
  Number of weeks retained in treatment based on a review of clinical records

SECONDARY OUTCOMES:
Completion of Substance Use Treatment | up to 12 weeks
  Treatment completed (yes or no) based on a review of clinical records
Days of Substance Use | up to 18 weeks
  Number of days of drug use based on self-report drug use and urine drug screen results
Days of Criminal Activity; Re-arrest; Incarceration | up to 18 weeks
  Number of crime days; re-arrest (yes or not); incarceration (yes or no) based on self-report information and public court record databases

OTHER OUTCOMES:
Rating of App Satisfaction | up to 12 weeks
  Rating of client satisfaction using the app based on self-report information

CONTACTS AND LOCATIONS:
Overall Officials: Steven B Carswell, Ph.D., Principal Investigator — COG Analytics
Locations (1):
- REACH Health Services, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
COG Analytics (COG) and Friends Research Institute (FRI) are committed to the open and timely dissemination of research outcomes. Investigators in the proposed study recognize that promising new methods, technologies, strategies and computer software may arise during the course of this research. The investigators are aware of, and agree to abide by, the principles for sharing research resources as described by the National Institutes of Health (NIH) in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources."